CLINICAL TRIAL: NCT01776229
Title: Exposure, Relaxation, & Rescripting Therapy-Child
Acronym: ERRT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Lisa Cromer, Associate Professor of Psychology, University of Tulsa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TU 11-63RI
Record Dates: First submitted 2012-07-24; First posted 2013-01-28 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Nightmares Associated With Trauma and Stress
Keywords: nightmare; PTSD; trauma; children; cognitive behavior therapy; stress; sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral (Experimental): Exposure, Relaxation, & Rescripting Therapy-Child utilizes behavioral and cognitive therapy techniques of exposure therapy and cognitive restructuring.
  Interventions: Behavioral: Exposure, Relaxation, & Rescripting Therapy-Child
- Waitlist Control (No Intervention): All potential participants will be evaluated and some will be randomly placed in the control group, following the five-week treatment phase, participants in the control group will be re-evaluated and offered the treatment

INTERVENTIONS:
Behavioral: Exposure, Relaxation, & Rescripting Therapy-Child — Exposure, Relaxation, & Rescripting Therapy (ERRT) will be conducted once a week for five consecutive weeks for approximately two hours per session. Each treatment session focuses on one of the following topics/skills: psycho-education and investment in treatment, psycho-education, Progressive Muscle Relaxation, diaphragmatic breathing,child-friendly exposure to the trauma-nightmare, and rescription.
  Arms: Behavioral

SUMMARY:
Untreated trauma-related nightmares and sleep-related disorders are associated with chronic health problems, burdening both the suffering individual and the health-care system. The study implements an innovative, cost-efficient, nightmare treatment for trauma-exposed children. It is the first randomized clinical trial with children, adapting an efficacious adult therapy to a 5-session nightmare treatment for 5-17 year-olds. Trauma nightmares are a mechanism in development and maintenance of secondary post-trauma psychopathology, medical problems and family dysfunction. Therefore, this treatment may prevent long-term secondary health and behavioral problems. It provides a viable healthcare option to Oklahomans, lessening long-term financial medical and behavioral health expenses. Scientific models currently view PTSD treatment as primary, often leaving nightmares untreated. That approach does not address the pernicious impact of trauma-nightmares in individuals with sub-threshold PTSD or whose nightmares are a primary condition. The theoretical innovation of this therapy can advance the field's understanding of the development of trauma sequelae.

ELIGIBILITY:
Inclusion Criteria:

* children age 5-17 with traumatic or potentially traumatic/adverse experiences and nightmares occurring at least once per week over a minimum of one month
* have a parent or legal guardian who is able to participate in treatment assignments at home and be able to read and speak English

Exclusion Criteria:

* adult, no traumatic experience, no nightmares, apparent psychosis, pervasive developmental disorder, or mental retardation, not able to read and speak English
* in order to ensure the verbal comprehension of the child, the PPVT will be used to help evaluate if a child is suitable for treatment, as an index to ensure they can verbally comprehend the cognitive component of treatment

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Trauma Related Nightmare Survey - Child Version (TRNS-C) Reflecting change in nightmare frequency, severity, and duration. | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The TRNS-C is a 14-item self-report measure that assesses current sleep quality, frequency, severity, and duration of nightmares, as well as cognitions, emotions, and behaviors related to nightmares in children.

SECONDARY OUTCOMES:
University of California at Los Angeles Post-traumatic Stress Disorder Reaction Index for the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) (UPID) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The UPID screens for trauma exposure and posttraumatic symptoms among youth 7 to 18 years old. Queries types of trauma exposures, assesses for DSM-IV criteria of traumatic exposure and the past-month frequency of PTSD symptoms and 2 associated features of PTSD in childhood.
Revised Child Anxiety and Depression Scale (RCADS) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The RCADS is a 47-item scale that corresponds to the DSM-IV anxiety disorders and it incorporates a sub scale for major depression. There is a six-factor structure with the following sub scales: Separation Anxiety Disorder, Social Phobia, Generalized Anxiety Disorder, Obsessive-Compulsive Disorder, Panic Disorder, and Major Depressive Disorder.
Nightmare Distress Questionnaire - Modified (NDQ) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The NDQ is a 13-item self-report measure of nightmare related distress. Higher scores are significantly related to interest in therapy for nightmares.
Pittsburgh Sleep Quality Index (PSQI) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The PSQI is a 19-item self-report measure of sleep quality and disturbance. It queries sleep quality and disturbances over the last month. Seven component scores are generated from this measure including: subjective sleep quality, latency, duration, habitual sleep efficiency, sleep problems, use of sleep medications, and daytime dysfunction.
Strengths and Difficulties Questionnaire - Child Version (SDQ) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The SDQ is a self-report instrument designed for completion by 11-16 year-olds. Specifically, children respond to 25 attributes (emotional, conduct, hyperactivity, peer relationships, and prosocial behaviors).
Child Behavior Checklist for Ages 6-18 (CBCL/6-18) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The CBCL can be completed by parents or parent-surrogates. It consists of 20 items that provide information regarding a child's competencies; 118 items assess both behavioral and emotional problems; and two open-ended questions for reporting additional problems.
Child Behavior Checklist for Ages 1.5-5 (CBCL/1.5-5) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The CBCL can be completed by parents or parent-surrogates. It consists of 99 items that assess both behavioral and emotional problems; and open-ended questions for reporting additional problems.
Children's Sleep Habits Questionnaire (CSHQ) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The CSHQ is a 33-item parent-report measure of sleep behavior that can be used by parents of children 4 to 12 years of age. A total score is derived from items from 8 sub scales: Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night Wakings, Parasomnias, Sleep-Disordered Breathing, and Daytime Sleepiness.
Strengths and Difficulties Questionnaire - Parent Version (SDQ) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The SDQ has two parent versions designed for 4-10 year-olds and 11-16 year-olds. Specifically, parents respond to 25 attributes (emotional, conduct, hyperactivity, peer relationships, and prosocial behavior).
The Parenting Stress Scale (PSS) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The PSS is an 18-item measure that assesses stress related to parenting (e.g., "I am happy in my role as a parent," "Having child(ren) has been a financial burden").
Pittsburgh Sleep Quality Index - Parent self-report (PSQI) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  Similar to the child version, the adult form of the PSQI is a 19-item self-report measure of sleep quality and disturbance. It queries sleep quality and disturbances over the last month. It will serve as an index of secondary gain from treatment by way of parent's improved sleep quality and quantity.
The McMaster Family Assessment Device (FAD) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The FAD is a 53-item measure that identifies seven dimensions of family functioning: Problem Solving, Communication, Roles, Affective Responses, Affective Involvement, Behavior Control, and General Functioning.
Behavior Rating Inventory of Executive Function - Parent Form (BRIEF) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The BRIEF is an 86-item measure that assesses different aspects of executive function behaviors in the home environment. There are eight different scales of executive function assessed within the measure.
Child Behavior Checklist - Teacher Form (CBCL-TR) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks.
  This form of the CBCL is to be completed by the child's teacher. It consists of 20 items that provide information regarding a child's competencies within school; 113 items that assess both behavioral and emotional problems; and one open-ended question for reporting additional problems.
Behavior Rating Inventory of Executive Function - Teacher Form (BRIEF) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks.
  The BRIEF is an 86-item measure that assesses different aspects of executive function behaviors in the school. There are eight different scales of executive function assessed within the measure.
Child Attention Network Task (Child ANT) | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  This is a computerized game that assesses attention. This measure presents a single fish or five fish in a horizontal row. Children are asked to respond to the center fish by pressing the left or right button on the computer mouse in the direction in which the fish is pointing.
Trail Making Test | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The Trail Making Test is a measure of visual attention and task switching. The test has two parts in which the child is instructed to connect a set of 25 dots as fast as possible while maintaining accuracy.
Animal Sorting | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  This subtest from the "A Developmental NEuroPSYchological Assessment" (NEPSY) assesses the ability to formulate basic concepts, to transfer those concepts into action, and to shift set from one concept to another.
Auditory Attention and Response Set | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  This subtest from the NEPSY has two parts. The Attention Auditory assesses selective auditory attention and the ability to sustain it. The Response Set assesses the ability to shift and maintain a new and complex set involving both inhibition of previously learned responses and correctly responding to matching or contrasting stimuli.
Clocks | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  This subtest from the NEPSY assesses planning and organization, visuoperceptual and visuospatial skills, and the concept of time related to analog clocks.
Actiwatch-2 Wrist Monitor | The wrist actigraph will be worn between session for a specified amount of time. The actigraph will be worn continously during the loan period except for swimming, other continous water sports, and bathing.
  This device is the size of a wristwatch. It records movement, which can be used to better understand sleep quality and sleep cycles. If also has a button for tracking nightmares. It is not a requirement of the study to wear the actigraph.
Letter-Number Sequencing | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  This subtest on the Wechsler Intelligence Scale for Children Fourth Edition (WISC-IV) assesses attention, short-term memory, and processing speed. The child will listen to a sequence of letters and numbers and then process, recall, repeat and manipulate these letters and numbers.
Digit span | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  This subtest of the WISC IV will be used to assess short-term memory, attention and concentration. The child participant will be asked to repeat numbers in the same order as read aloud by the examiner and in reverse order as read by the examiner.
R-CBM | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The Reading Curriculum Based Measurement of the Aimsweb reading system will be used as a measure of a child's oral reading skill and speed. This measure was designed to assess general reading achievement and comprehension. For each administration of an R-CBM probe, the child will read a passage aloud for one minute. Words that are mispronounced, substituted, omitted or read out of sequence that the child does not self-correct within three seconds are to be recorded as errors.
MAZE | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for followups at 3 months and 6 months post treatment.
  The Standard Reading Comprehension Assessment Passages (MAZE-CBM) subtest of the Aimsweb Measurement System will be used in conjunction with the R-CBM, as a supplemental measure to provide a more complete picture of the child's general reading skill and speed. This measure was designed to corroborate a child's general reading achievement and comprehension score of the R-CBM. The MAZE probe is a multiple choice cloze task that the child reads silently. The first sentence of a 150-400 word paragraph is left intact. Thereafter, every seventh word is replaced with three words inside parentheses and the child will choose the word that correctly completed the sentence.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cromer, Phd, Principal Investigator — The University of Tulsa
Locations (1):
- The University of Tulsa Institute for Trauma Abuse and Neglect, Tulsa, Oklahoma, United States

REFERENCES:
- See also: Child Nightmare Study Facebook Information Page — https://www.facebook.com/ChildNightmareStudy